CLINICAL TRIAL: NCT04899999
Title: Graphic Messages to Prevent E-Cigarette Use Among Latino and African American Adolescents: A Randomized Controlled Trial
Brief Title: Graphic Messages to Prevent E-Cigarette Use Among Black and Latino Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Francisco Cartujano, MD, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006267; U54CA228110 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2022-02

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Financial reward graphic message (Experimental)
  Interventions: Behavioral: Financial reward graphic message
- Health reward graphic message (Experimental)
  Interventions: Behavioral: Health reward graphic message
- Self-efficacy graphic message (Experimental)
  Interventions: Behavioral: Self-efficacy graphic message
- Social norms graphic message (Experimental)
  Interventions: Behavioral: Social norms graphic message

INTERVENTIONS:
Behavioral: Financial reward graphic message — Graphic image will be shared with the participants online once in either English or Spanish depending on their language of preference. Image includes the following text: Vaping leads to nothing. Don't let your money vaporize away.
  Arms: Financial reward graphic message
Behavioral: Health reward graphic message — Graphic image will be shared with the participants online once in either English or Spanish depending on their language of preference. Image includes the following text: Dying for a vape? It hurts more than you know.
  Arms: Health reward graphic message
Behavioral: Self-efficacy graphic message — Graphic image will be shared with the participants online once in either English or Spanish depending on their language of preference. Image includes the following text: Vaping companies are targeting Black and Latino teens. Your life matters. Don't let them take it away.
  Arms: Self-efficacy graphic message
Behavioral: Social norms graphic message — Graphic image will be shared with the participants online once in either English or Spanish depending on their language of preference. Image includes the following text: Just because vaping is common, doesn't mean it's cool. Stay woke. Don't smoke.
  Arms: Social norms graphic message

SUMMARY:
The aim of this study is to determine if graphic messages prevent future vaping use among African American and Latino adolescents. The images have been developed in a user-design model and include four main themes: health reward, financial reward, self-efficacy, and social norms. We will assess pre- and post-exposure reactions on likelihood of future vaping among African American and Latino adolescents.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American/Black and/or Hispanic/Latino
* know how to read and speak English and/or Spanish
* have never used e-cigarettes
* have access to a device that will be able to connect to the online survey

Exclusion Criteria:

* not identifying as African American/Black and/or Hispanic/Latino
* using e-cigarettes

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message
Started | 93 | 88 | 92 | 89
Completed | 93 | 88 | 92 | 89
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message | Total
Number analyzed (Participants) | 93 | 88 | 92 | 89 | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.04 (1.61) | 15.06 (1.35) | 15.00 (1.46) | 14.89 (1.52) | 15.00 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 person in each of the financial rewards, self-efficacy and social norms arms reported as transgender.
  Participants
    number analyzed (Participants) | 92 | 88 | 91 | 88 | 359
    Female | 38 | 34 | 26 | 26 | 124
    Male | 54 | 54 | 65 | 62 | 235
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 45 | 46 | 46 | 44 | 181
  Black/African American | 48 | 42 | 46 | 45 | 181
Region of Enrollment [Number; unit: participants]
  United States | 89 | 81 | 86 | 88 | 344
  Puerto Rico | 4 | 7 | 6 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Participants Susceptible to Future Vaping
Description: Susceptibility to future vaping was assessed before and after exposure to the graphic messages. Informed by prior foundational research on youth electronic cigarette use, susceptibility was measured with three items assessing curiosity, intent, and social influence. Participants were asked, "Have you ever been curious about using e-cigarettes/vaping?", "Do you think that you will use e-cigarettes/vape in the next 12 months?", and "If one of your best friends were to offer you an e-cigarette/electronic vapor product, would you use it?" (1 = "Definitely not" to 4 = "Definitely yes"). Responses were dichotomized: participants were categorized as susceptible if they answered anything other than "Definitely not" to at least one item. The percentage of susceptible participants was calculated before and after exposure; change in percentage reflects the difference.
Time Frame: baseline to post-intervention, approximately 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message
Number analyzed (Participants) | 93 | 88 | 92 | 89
percentage of participants | 1.1 | -5.7 | -2.3 | -3.2

2. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied With the Graphic Message
Description: Satisfaction with the assigned vaping prevention graphic message was assessed using the item: "How satisfied are you with the image?" Responses were recorded on a 5-point Likert scale from 1 = "Extremely unsatisfied" to 5 = "Extremely satisfied." Participants selecting 5 ("Extremely satisfied") were categorized as satisfied. The percentage of satisfied participants was calculated per group. Higher percentages indicate greater satisfaction with the message.
Time Frame: Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message
Number analyzed (Participants) | 93 | 88 | 92 | 89
percentage of participants | 68.8 | 69.3 | 34.7 | 56.1

3. Secondary Outcome: Percent of Participants Who Would Recommend the Graphic Message to a Friend
Description: participants were asked, "Would you recommend this picture to a friend?" with response options of Yes or No. The percentage of participants who responded "Yes" was calculated per group. Higher percentages indicate greater endorsement of the message.
Time Frame: Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message
Number analyzed (Participants) | 93 | 88 | 92 | 89
percentage of participants | 90.3 | 94.3 | 70.6 | 80.8

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Financial Reward Graphic Message | Health Reward Graphic Message | Self-efficacy Graphic Message | Social Norms Graphic Message
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/88 | 0/92 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/88 | 0/92 | 0/89
Other Adverse Events (participants affected / at risk) | 0/93 | 0/88 | 0/92 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04899999/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04899999/ICF_001.pdf